CLINICAL TRIAL: NCT07299253
Title: Preclinical Safety Evaluation and First-in-Human Translational Study of [177Lu]Lu-TEFAPI-06: A Novel Albumin-Binding FAPI Radiopharmaceutical for Theranostics
Brief Title: Preclinical Safety Evaluation and First-in-Human Translational Study of [177Lu]Lu-TEFAPI-06
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lanzhou University Second Hospital (Other)
Responsible Party: Principal Investigator, Jiangyan Liu, Director of the Nuclear Medicine Department of the Second Hospital of Lanzhou University, Lanzhou University Second Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023A-371
Record Dates: First submitted 2025-11-26; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Solid Tumors (Any Localization)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with advanced metastatic solid tumors (Experimental)
  Interventions: Drug: radionuclide therapy with [177Lu]Lu--TEFAPI-06

INTERVENTIONS:
Drug: radionuclide therapy with [177Lu]Lu--TEFAPI-06 — A Novel Albumin-Binding FAPI Radiopharmaceutical for Theranostics

SUMMARY:
This study aims to systematically evaluate the safety, biodistribution, dosimetry, and preliminary therapeutic potential of [177Lu]Lu-TEFAPI-06 through an exploratory first-in-human (FIH) trial.

DETAILED DESCRIPTION:
This study represents a comprehensive "bench-to-bedside" translational investigation, providing the first systematic report on the safety profile of [177Lu]Lu-TEFAPI-06-a novel albumin-binding fibroblast activation protein inhibitor (FAPI) radiopharmaceutical-and its successful transition into a FIH. The investigators preliminarily evaluated its safety, dosimetry, and therapeutic response in patients with ibroblast activation protein (FAP)-overexpressing metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically confirmed advanced metastatic solid tumors refractory or intolerant to standard therapies
* ECOG performance status 0-2
* Life expectancy > 3 months
* At least one FAP-avid lesion confirmed by baseline [18F]-FAPI PET/CT
* Adequate organ and bone marrow function prior to the first dose

Exclusion Criteria:

* Chemotherapy, radiotherapy, or targeted therapy within 4 weeks
* Severe hepatic or renal dysfunction
* Uncontrolled active infection or severe comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2025-08-16 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Treatment-Emergent Adverse Events (TEAEs) as Assessed by CTCAE v5.0 | From Baseline up to 30 days after the last dose of study intervention (approximately 4 weeks)
  Safety and tolerability will be assessed by recording the frequency, duration, and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs). The assessment includes clinically significant changes in vital signs (blood pressure, heart rate, respiratory rate, temperature), physical examination findings, 12-lead Electrocardiogram (ECG) parameters, and clinical laboratory tests (including Complete Blood Count [CBC], Urinalysis, Liver Function Tests [LFTs], and Renal Function Tests). Severity of adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0.

SECONDARY OUTCOMES:
Change from Baseline in [18F]-FAPI PET/CT Parameters in Target Lesions | Baseline (Day 0) and 1 month post-treatment.
  [18F]-FAPI PET/CT images will be acquired to evaluate the expression of FAP within the tumor stroma. The efficacy assessment will be based on the quantitative analysis of Standardized Uptake Values (SUVmax and SUVmean) and Tumor-to-Background Ratios (TBR) of the target lesions. Changes in tracer uptake between the baseline scan and the follow-up scan will be calculated.
Change from Baseline in Tumor-Specific Serum Marker Levels | Baseline (Day 0) and 1 month post-treatment.
  Peripheral blood samples will be collected to measure the serum concentration of tumor-specific biomarkers relevant to the indication (e.g., CEA, CA19-9, PSA, or other applicable markers). The change in concentration levels will be assessed to evaluate biochemical response.

OTHER OUTCOMES:
Biodistribution and Pharmacokinetics of [177Lu]Lu-TEFAPI-06 | 0.5, 2, 24, 48, 72, and 120 hours post-injection.
  Biodistribution will be assessed by quantitative analysis of Whole-Body planar and SPECT/CT images. Tracer uptake in blood, normal organs (kidneys, liver, etc.), and tumor tissues will be quantified at serial time points. Parameters to be analyzed include the percentage of injected dose (%ID) and percentage of injected dose per gram (%ID/g) for each regions of Interest (ROI) .
Radiation Absorbed Doses in Normal Organs and Tumor Lesions | Post-injection at 0.5, 2, 24, 48, 72, and 120 hours.
  Radiation dosimetry will be calculated based on biodistribution data derived from serial imaging. Following the administration of [177Lu]Lu-TEFAPI-06, Whole-Body (WB) planar scintigraphy and SPECT/CT scans will be performed. ROIs will be drawn over source organs and tumor lesions to generate time-activity curves. Absorbed doses (in Gy/GBq) will be estimated using standard dosimetry software (e.g., OLINDA/EXM or IDAC) based on the MIRD scheme.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital & Clinical Medical School, Lanzhou University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT07299253/Prot_SAP_000.pdf